CLINICAL TRIAL: NCT03190551
Title: A Randomized Controlled Trial Comparing Retroclavicular and Costoclavicular Approach for Infraclavicular Brachial Plexus Block
Brief Title: Retroclavicular Versus Costoclavicular Approach for Infraclavicular Brachial Plexus Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AntalyaTRH15
Record Dates: First submitted 2017-06-12; First posted 2017-06-19 (Actual); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Disorder of Upper Extremity
Keywords: infraclavicular brachial plexus block; retroclavicular approach; costoclavicular approach; upper limb surgery; needle shaft visibility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- retroclavicular approach (Active Comparator): Patients in this group will be randomized to receive an retroclavicular approach to Ultrasound Guided Infraclavicular Brachial Plexus Nerve Block .
  Interventions: Other: retroclavicular approach
- costoclavicular approach (Active Comparator): Patients in this group will be randomized to receive an costoclavicular approach to Ultrasound Guided Infraclavicular Brachial Plexus Nerve Block .
  Interventions: Other: costoclavicular approach

INTERVENTIONS:
Other: retroclavicular approach — Retroclavicular approach for ultrasound guided infraclavicular brachial plexus block
  Arms: retroclavicular approach
Other: costoclavicular approach — costoclavicular approach for ultrasound guided infraclavicular brachial plexus block
  Arms: costoclavicular approach

SUMMARY:
The primary aim of this study is to compare needle shaft visibility between the retroclavicular approach and costoclavicular approach for infraclavicular brachial plexus block in patients undergoing elective upper limb surgery. Secondary aim is to investigate the differences between the two groups in sensorial block success rate, block performance time, block performance related pain, motor block success rate, surgical success rate, complications, patient satisfaction, use of supplemental local anesthetic, use of analgesic.

DETAILED DESCRIPTION:
Infraclavicular blocks are performed with different approaches. This study evaluated the effectiveness, safety and feasibility of a retroclavicular brachial plexus block as compared with costoclavicular approach for infraclavicular brachial plexus block. 60 patients scheduled for elective upper limb surgery were recruited and randomized into two groups: Retroclavicular approach for infraclavicular block (Group I), costoclavicular approach for infraclavicular block (Group R). Sensory block, adverse effects and complications were evaluated and recorded every 5 minutes until 30 min after local anesthetic injection. Success rate of each nerve sensory block, complications, rate of satisfaction, rate of failure and incidence rate of adverse effects, the needle shaft visibility, procedure time,duration of the block's effect, use of supplemental local anesthetic, use of analgesic are compared with both groups.

ELIGIBILITY:
Inclusion Criteria:

* patients who undergo elective forearm or hand surgery under infraclavicular brachial plexus block
* American Society of Anesthesiologists class 1 to 3
* Ability to consent

Exclusion Criteria:

* History of allergic reaction to local anaesthetics
* Peripheral neuropathy
* Renal or hepatic insufficiency
* Coagulation disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Needle shaft visibility | 10 minutes after the needle inserted the skin
  Needle visibility reviewed by two anesthesiologists using a 5-point Likert scale

SECONDARY OUTCOMES:
Technique duration | Time required in seconds for the block completion (10 minutes)
  Number of seconds needed to complete the block, from time of local skin anesthesia until regional block needle removal.
Patient satisfaction using a visual analogue scale | Assessed 24 hours after the block
  Using a visual analog scala, patients will quantify their satisfaction with the retroclavicular and costaclavicular technique .
supplemental analgesic used | 90 minutes after block completion
  The use of supplementary local anesthetic and the use of intravenous narcotics were recorded.
complications such as pneumothorax, hemothorax, intraarterial injection, intravenous injection | 24 hours
  Asked about possible complications
motor block success rate | Assessed 40 minutes after block completion
  Success is defined as complete motor block in the distribution of the radial, median, ulnar, musculocutaneous nerves of the forearm and hand
Success Rate of the sensorial Block | Assessed 30 minutes after block completion
  Success is defined as complete sensory loss in the distribution of the radial, median, ulnar, musculocutaneous, and medial cutaneous nerves of the forearm and hand
Block performance related pain | 10 minutes after the needle inserted the skin
  Block performance related pain was evaluated with a visual analog scala after the removal of the needle.

CONTACTS AND LOCATIONS:
Overall Officials: Hayri Fatih Metinyurt, MD, Study Director — Antalya Training and Research Hospital; Nilgun Kavrut Ozturk, MD, Principal Investigator — Antalya Training and Research Hospital; Ali Sait Kavakli, MD, Principal Investigator — Antalya Training and Research Hospital
Locations (1):
- Antalya Training and Research Hospital, Department of Anesthesiology and Reanimation, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No